CLINICAL TRIAL: NCT07401810
Title: The Effect of Facial Yoga Practice on Perceived Stress, Cognitive Control, Cognitive Flexibility, and Cortisol Levels in Menopausal Women
Brief Title: Facial Yoga in Menopausal Women
Acronym: FacialYogaM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Ayşe Eminoğlu, Research Assistant, Marmara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MU-SBF-ETIK-206
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Menopause; Stress, Psychological; Cortisol; Cognitive Flexibility; Nonpharmacological Interventions; Randomized Controlled Trial; Cognitive Control; Perceived Stress; Yoga
Keywords: Menopause; Perceived Stress; Cognitive Flexibility; Cognitive Control; Yoga; Cortisol; Saliva
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Facial Yoga Intervention (Experimental)
  Interventions: Behavioral: Facial Yoga Program
- Usual Care (No Intervention)

INTERVENTIONS:
Behavioral: Facial Yoga Program — A structured 12-week online facial yoga program consisting of two 60-minute sessions per week. The intervention focuses on facial myofascial relaxation, breathing regulation, and body awareness for stress regulation and cognitive functioning. Sessions will be conducted in a group format, and no audio or video recordings will be taken.
  Arms: Facial Yoga Intervention

SUMMARY:
Purpose: The purpose of this study is to evaluate the effects of a structured facial yoga-based behavioral intervention on perceived stress, cognitive control, cognitive flexibility, and salivary cortisol levels in women during the menopausal period. The study aims to determine whether a non-pharmacological and non-invasive behavioral intervention can support psychological and cognitive functioning and reduce biological stress responses in menopausal women.

Design: This study is designed as a randomized, controlled, pretest-posttest experimental trial with a post-intervention follow-up assessment. Eligible participants will be randomly assigned to either an intervention group or a control (usual care) group. Outcomes will be assessed at baseline, immediately after the intervention, and at follow-up to evaluate both the immediate and sustained effects of the intervention.

Method: A total of 100 menopausal women aged 45-65 years will be recruited from a menopause outpatient clinic and randomly allocated to either the intervention group or the control group. The intervention group will participate in a 12-week online facial yoga program consisting of two 60-minute sessions per week.

In this study, facial yoga refers to a non-pharmacological and non-invasive behavioral intervention focusing on facial myofascial relaxation, breathing regulation, and body awareness for stress regulation and cognitive functioning. The program will include facial myofascial relaxation techniques, basic yoga postures suitable for all physical levels, and structured breathing exercises. All sessions will be conducted online in a group format, and no audio or video recordings will be taken.

The control group will continue to receive routine outpatient care during the study period and will be offered the facial yoga program after the completion of follow-up assessments, upon request.

Data will be collected at three time points: at baseline prior to the intervention, immediately after completion of the 12-week intervention, and at 8 weeks following the intervention as a follow-up assessment. Perceived stress, cognitive control, and cognitive flexibility will be assessed using validated self-report questionnaires. Salivary cortisol samples will be collected under standardized morning conditions at each assessment point to evaluate biological stress response.

Hypotheses:

H1: Menopausal women participating in the facial yoga intervention will demonstrate a significant reduction in perceived stress levels compared to the control group at post-intervention and follow-up assessments.

H2: Menopausal women participating in the facial yoga intervention will demonstrate a significant reduction in salivary cortisol levels compared to the control group at post-intervention and follow-up assessments.

H3: Menopausal women participating in the facial yoga intervention will demonstrate a significant improvement in cognitive control and cognitive flexibility compared to the control group at post-intervention and follow-up assessments.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged 45-65 years
* In the menopausal period, defined as at least 12 months since the last menstrual period
* Able to read and understand Turkish and to complete self-report questionnaires

Exclusion Criteria:

* Current or past diagnosis of a psychiatric disorder or ongoing psychiatric treatment
* Regular use of antidepressant, anxiolytic, or corticosteroid medications
* History of cancer or currently receiving active oncological treatment
* Participation in facial yoga or similar yoga-based programs within the past 6 months
* Any medical condition that may prevent safe participation in mild physical activity
* Incomplete attendance to intervention sessions or incomplete outcome data during the study period

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is gender-based because it focuses exclusively on women in the menopausal period, a biological condition that occurs only in females. Eligibility criteria are therefore limited to female participants.
Enrollment: 100 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress Level | Baseline, immediately post-intervention (12 weeks), and 8 weeks post-intervention follow-up
  Change in perceived stress levels measured using the Perceived Stress Scale (PSS-14). The scale consists of 14 items rated on a 5-point Likert scale (0-4), with total scores ranging from 0 to 56. Higher scores indicate higher perceived stress levels.
Salivary Cortisol Level | Baseline, immediately post-intervention (12 weeks), and 8 weeks post-intervention follow-up
  Change in salivary cortisol levels measured from morning saliva samples collected under standardized conditions.
Cognitive Control and Flexibility | Baseline, immediately post-intervention (12 weeks), and 8 weeks post-intervention follow-up
  Change in cognitive control and cognitive flexibility levels measured using the Cognitive Control and Flexibility Questionnaire. The questionnaire consists of two subscales (cognitive control and cognitive flexibility), with items rated on a 7-point Likert scale. Higher scores indicate better cognitive control and greater cognitive flexibility.

IPD SHARING:
Plan to Share IPD: No